CLINICAL TRIAL: NCT00785343
Title: Effectiveness of Adding Robotic Therapy to Conventional Therapy for Acute Stroke Patients With Upper Extremity Paresis
Brief Title: Study of Robot-assisted Arm Therapy for Acute Stroke Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Kevin Terry, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-618-08
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Acute Stroke; Paresis
Keywords: stroke; acute; arm; robot; therapy; arm paresis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Treatment (Active Comparator)
  Interventions: Procedure: Conventional Therapy
- Robotic and Conventional Therapy (Experimental)
  Interventions: Device: Reo Go robotic arm trainer

INTERVENTIONS:
Device: Reo Go robotic arm trainer — Robotic training with the Reo Go is included with conventional treatment during daily OT sessions
  Arms: Robotic and Conventional Therapy
Procedure: Conventional Therapy — Occupational therapy that is the current standard of care
  Arms: Conventional Treatment

SUMMARY:
The purpose of this study is to compare standard occupational therapy to a combination of conventional (standard) and robotic therapy. The Reo Go device will provide robotic therapy that gives therapists a tool that could make stroke treatment faster and better by helping patients practice more accurate arm movements with help from the device.

DETAILED DESCRIPTION:
HYPOTHESES

* Motor function will be significantly greater for the patients in the robotic training group as measured by standard clinical evaluations.
* Functional independence gains will be similar for both groups because the robotic therapy is not task-specific for activities of daily living (ADL).
* Robotic training will reduce pain and spasticity more effectively than conventional therapy alone, due to increased number of movements performed during the robotic training.
* Muscle activation patterns for patients receiving robotic training will show decreased agonist/antagonist co-contraction and less erratic muscle activation.
* Robotic training patients will demonstrate significantly greater ROM, movement accuracy and higher movement speed during exercises performed as part of robotic training. For robotic exercises performed only as part of the robotic assessment, these improvements will be significantly less than those for practiced movements.

ELIGIBILITY:
Inclusion criteria Right hemisphere, unilateral ischemic stroke with onset of less than 15 days that results in arm weakness Right-handed 65-84 years of age Manual Muscle Test score of at least 2/5 Must be able to follow 2-3 step commands Head, neck, and trunk control to maintain an upright posture for a minimum of 45 minutes Some synergistic movement at shoulder Active shoulder flexion and/or abduction greater then 30 degrees Active elbow flexion of 45 degrees or more

Exclusion criteria

* Previous stroke history
* Hemorrhagic stroke, cerebellar stroke, or subarachnoid hemorrhage
* Contractures in the involved upper extremity at the shoulder, elbow, or wrist
* Moderate to severe tone in the involved upper extremity
* Flaccid involved upper extremity
* Full, active isolated movement of the involved upper extremity
* Corrected visual acuity worse than 20/50 for distance
* Cognitive or other deficits that would negatively affect their ability to follow directions or track visual targets
* Unstable cardiovascular orthopedic or neurological conditions that would preclude exercise in short-duration, high work-load trials

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-09

PRIMARY OUTCOMES:
Fugl-Meyer Score | Start and end of treatment

SECONDARY OUTCOMES:
EMG - muscle activation and co-contraction index | Start and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lauren McDonagh, PT, Principal Investigator — Kessler Rehabilitation Institute
Locations (1):
- Kessler Institute for Rehabilitation, Saddle Brook, New Jersey, United States

REFERENCES:
- [Background] Lum PS, Burgar CG, Shor PC. Evidence for strength imbalances as a significant contributor to abnormal synergies in hemiparetic subjects. Muscle Nerve. 2003 Feb;27(2):211-21. doi: 10.1002/mus.10305. PMID 12548529
- [Background] Prange GB, Jannink MJ, Groothuis-Oudshoorn CG, Hermens HJ, Ijzerman MJ. Systematic review of the effect of robot-aided therapy on recovery of the hemiparetic arm after stroke. J Rehabil Res Dev. 2006 Mar-Apr;43(2):171-84. doi: 10.1682/jrrd.2005.04.0076. PMID 16847784